CLINICAL TRIAL: NCT03098706
Title: Impact of Therapeutic Hypothermia in Expanded Criteria Brain-dead Donors on Kidney-graft Function in the Kidney-transplant Recipients: Multicenter Randomized Controlled Trial" HYPOREME
Brief Title: Therapeutic Hypothermia in "Expanded Criteria" Brain-dead Donors and Kidney-graft Function
Acronym: HYPOREME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RC16_0041
Record Dates: First submitted 2017-02-15; First posted 2017-04-04 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Organ Donor; Brain Death; Kidney Transplant; Complications; Critical Illness; Hypothermia
MeSH Terms: conditions — Brain Death; Critical Illness; Hypothermia | interventions — Hypothermia, Induced

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NT normothermia (Other): After information for donation and research has been explained, organ donors in the normothermia (NT) group will either be maintained to spontaneously reach a body temperature of 36,5 °C-37,5°, until transfer to the operating room.
  Interventions: Procedure: Procedure control: normothermia
- HT mild hypothermia (Experimental): The intervention will take place after information for donation and research has been explained . Organ donors in the intervention group will either be actively warmed or allowed to reach a body temperature of 34 °C-35°C, until transfer to the operating room.
  Interventions: Procedure: Procedure active

INTERVENTIONS:
Procedure: Procedure control: normothermia — Temperature will be maintained between 36.5° and 37.5°C in the control group. In case of temperature superior to 37.5°C or inferior to 36.5°C, a pharmaceutical treatment and/or active cooling or warming will be introduce to maintain temperature between the range of 36.5 - 37.5°C.
  Other Names: Normothermia
  Arms: NT normothermia
Procedure: Procedure active — Therapeutic hypothermia ie targeted controlled temperature between 34° and 35°C will be induced in the active group. Usual method of controlled temperature will be used in ICU: internal active method or external active method.
  Other Names: Therapeutic hypothermia/ Induce hypothermia
  Arms: HT mild hypothermia

SUMMARY:
Each year, only one third of patients registered on the waiting list receive a kidney transplant. Numerous paths are being explored with the aim of reversing this shortage. The first is to increase the number of organs by developing harvesting from donors in a state of brain-death (BD) termed "expanded criteria donors" or from patients deceased from circulatory arrest.

Another fundamental factor is to insure the success of the transplant by limiting the dysfunction of donor kidneys, marked by a delayed graft function (DFG).

The development of techniques to insure correct perfusion of harvested organs, and the optimization of reanimation and intensive care of brain-dead donors constitute important factors in DGF reduction.

Therapeutic Hypothermia could to be an attractive care strategy for BD patients.

ELIGIBILITY:
Inclusion Criteria:

* For donors: legal determination of death by neurologic criteria/deceased organ donor/no medical contre-indication to donation/Information given to the authorizing surrogate/ Pregnant women.

  * For transplant recipients : age 18 years or greater /information given and no opposition signed by recipients.

Exclusion Criteria:

* For donors: no legal determination of death by neurologic criteria/not a deceased organ donor/ medical contre-indication to donation/ no Information given to the authorizing surrogate.
* For transplant recipients: age <18 years / no information given and/or opposition signed by recipients.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
rate of patients with delayed graft function (DGF) | Day 7
  DGF is the recipient's requirement for dialysis during the first week after transplantation.
  To show the interest of Targeted Temperature Management in order to optimize the functional recovery of transplanted kidney transplants by comparing 2 groups of recipient subjects: those receiving one Graft from an "expanded criteria donors" maintained in hypothermia (34°-35°) and those receiving a graft from an "expanded criteria donors" maintained in normothermia (36,5°-37,5°).

SECONDARY OUTCOMES:
Temperature Profile | 24 hours
  comparison of temperature profile between the two arms
Severe arrhythmias | 24 hours
  Severe arrythmia will be define by salvo of ventricular extrasystole, ventricular fibrillation, ventricular tachycardia, need an external shock, need anti-arrhythmic treatment. Participants will be followed for the duration of Intensive Care Unit stay and/or operating room, an expected average of 24 hours.
Cardiac arrest | 24 hours
  SParticipants will be followed for the duration of Intensive Care Unit stay and/or operating room, an expected average of 24 hours.
Occurrence of hypotension measured by Total dose of inotropic drugs | 24 hours
  Total dose of different inotropic drugs (Epinephrine, Norepinephrine, Dobutamine) will be compare between 2 groups during targetted controlled temperature management period.
Occurrence of hypotension measured by cumulative fluid balance | 24 hours
  Cumulative fluid balance will be compare between 2 groups during targetted controlled temperature management period
occurrence of cardiac arrest | 24 hours
  comparison of occurrence of cardiac arrest between the two arms
Kidney function measured by serum creatinine value | 24 hours
  Kidney function measured by serum creatinine value
Kidney function measured by CKD EPI score | 24 hours
  Kidney function measured by CKD EPI score (= 141 x min(Scr/K,1)a x max(Scr/K,1)-1,209 x 0,993Age x 1,018 (for women))
electrolyte balance : potassium, calcium, sodium concentration disorders in mmoL/L | 24hours
  Potential hypothermia related side effects
glycemia in mmoL/L | 24hours
  Potential hypothermia related side effects
liver disorder (ASAT, ALAT, GGT, PAL , BILI in UI/L ) | 24hours
  Potential hypothermia related side effects
thrombocytopenia in mm3/L | 24hours
  Potential hypothermia related side effects
Number of individual organs transplanted | 24 hours
  Participants will be followed for the duration of Intensive care unit length of stay, and operating room, an average of 24 hours.
Hospital mortality | Day 7
  Participants will be followed for the duration of hospital stay, an expected average of 1 week.
Kidney function measured by serum creatinine value | Day 7
  Kidney function measured by serum creatinine value at day7
Kidney function measured by CKD EPI | Day 7
  Kidney function measured by CKD EPI (= 141 x min(Scr/K,1)a x max(Scr/K,1)-1,209 x 0,993Age x 1,018 (for women))
Extra renal support requirement | Day 7
  Extra renal support requirement at Day7
Kidney graft acute rejection | Day 7
  Kidney graft acute rejection
Acute pulmonary oedema by left ventricular failure | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days.
Severe arrythmia | Day 7
  Severe arrythmia will be define by salvo of ventricular extrasystole, ventricular fibrillation, ventricular tachycardia, need an external shock, need anti-arrhythmic treatment.
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Pulmonary embolism | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Acute coronary syndrome | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Nosocomial Bloodstream infection | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Early onset pneumonia | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Central Venous Catheter infection | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Urinary tract sepsis | Day 7
  Participants will be followed for the duration of transplantation unit stay, an expected average of 7 days
Mortality at D28 | D28
  comparison of mortality at D28 between the two arms
Mortality at 3 months | 3 months
  comparison of mortality at 3months between the two arms
Mortality at 1 year | 1 year
  comparison of mortality at 1 year between the two arms
Length of hospital stay | 48months
  comparison of length of hospital stay between the two arms
Kidney function measured by serum creatinine value | D28
  Kidney function measured by serum creatinine value
Kidney function measured by CKD EPI | D28
  Kidney function measured by CKD EPI (= 141 x min(Scr/K,1)a x max(Scr/K,1)-1,209 x 0,993Age x 1,018 (for women)) at Day28
Extra renal support requirement defined by percentage of patients requiring at least one dialysis | D28
  Extra renal support requirement
Kidney graft acute rejection | D28
  Kidney graft acute rejection
Acute pulmonary oedema by left ventricular failure | D28
  Acute pulmonary oedema by left ventricular failure
Severe arrythmia | D28
  Severe arrythmia will be define by salvo of ventricular extrasystole, ventricular fibrillation, ventricular tachycardia, need an external shock, need anti-arrhythmic treatment.
Pulmonary embolism | D28
  Pulmonary embolism
Acute coronary syndrome | D28
  Acute coronary syndrome
Nosocomial Bloodstream infection | D28
  Nosocomial Bloodstream infection
Early onset pneumonia | D28
  Early onset pneumonia
Central Venous Catheter infection | D28
  Central Venous Catheter infection
Urinary tract sepsis | D28
  Urinary tract sepsis
Kidney function measured by serum creatinine value | 3 months
  Kidney function measured by serum creatinine value
Kidney function measured by CKD EPI | 3 months
  Kidney function measured by CKD EPI (= 141 x min(Scr/K,1)a x max(Scr/K,1)-1,209 x 0,993Age x 1,018 (for women))
Extra renal support requirement defined by percentage of patients requiring at least one dialysis | 3 months
  Extra renal support requirement
Kidney function measured by serum creatinine value | 12 months
  Kidney function measured by serum creatinine value
Kidney function measured by CKD EPI | 12 months
  Kidney function measured by CKD EPI (= 141 x min(Scr/K,1)a x max(Scr/K,1)-1,209 x 0,993Age x 1,018 (for women))
Extra renal support requirement defined by percentage of patients requiring at least one dialysis | 12 months
  Extra renal support requirement

CONTACTS AND LOCATIONS:
Locations (54):
- France (54):
  - CHU Amiens-Picardie, Amiens
  - CHU d'Angers, Angers
  - CH Angouleme, Angoulême
  - CH Avignon, Avignon
  - CH de Blois, Blois
  - CHU de Bordeaux, Bordeaux
  - CH Bourges, Bourges
  - CHU Brest, Brest
  - CHU Caen, Caen
  - Ch Cholet, Cholet
  - Chu Clermont Ferrand, Clermont-Ferrand
  - Hopital Henri Mondor, Créteil
  - CHU de Dijon, Dijon
  - CH de Dreux, Dreux
  - CHU Grenoble, Grenoble
  - CH Marne la Vallée (GHEF), Jossigny
  - CH La Roche sur Yon, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CH Laval, Laval
  - Hopital Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CH Lorient, Lorient
  - CHU de Lyon, Lyon
  - Hopital de la Conception, Marseille
  - Hopital de la Timone, Marseille
  - CH de Meaux (GHEF), Meaux
  - CHU Montpellier, Montpellier
  - CH Morlaix, Morlaix
  - Nantes University Hospital, Nantes
  - CHU Nice, Nice
  - CH Orléans, Orléans
  - Hopital Saint Louis, Paris
  - Hopital de la Pitié Salpetriere, Paris
  - Hopital Necker, Paris
  - CHU Tenon, Paris
  - CHU Poitiers, Poitiers
  - CH Annecy Genevois, Pringy
  - CH Cornouaille, Quimper
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CH Saint Brieuc, Saint-Brieuc
  - CHRU Saint-Etienne, Saint-Etienne
  - CH Saint Nazaire, Saint-Nazaire
  - CH Saintes, Saintes
  - CH Saint Malo, St-Malo
  - CHU Strasbourg, Strasbourg
  - CHU Foch, Suresnes
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - CH Vannes, Vannes

REFERENCES:
- [Derived] HYPOREME Trial Group. Hypothermia for expanded criteria organ donors in kidney transplantation in France (HYPOREME): a multicentre, randomised controlled trial. Lancet Respir Med. 2024 Sep;12(9):693-702. doi: 10.1016/S2213-2600(24)00117-6. Epub 2024 Jun 11. PMID 38876137
- [Derived] Brule N, Canet E, Pere M, Feuillet F, Hourmant M, Asehnoune K, Rozec B, Duveau A, Dube L, Pierrot M, Humbert S, Tirot P, Boyer JM, Martin-Lefevre L, Labadie F, Robert R, Benard T, Kerforne T, Thierry A, Lesieur O, Vincent JF, Lesouhaitier M, Larmet R, Vigneau C, Goepp A, Bouju P, Quentin C, Egreteau PY, Huet O, Renault A, Le Meur Y, Venhard JC, Buchler M, Michel O, Voellmy MH, Herve F, Schnell D, Courte A, Glotz D, Amrouche L, Hazzan M, Kamar N, Moal V, Bourenne J, Le Quintrec-Donnette M, Morelon E, Boulain T, Grimbert P, Heng AE, Merville P, Garin A, Hiesse C, Fermier B, Mousson C, Guyot-Colosio C, Bouvier N, Rerolle JP, Durrbach A, Drouin S, Caillard S, Frimat L, Girerd S, Albano L, Rostaing L, Bertrand D, Hertig A, Westeel PF, Montini F, Delpierre E, Dorez D, Alamartine E, Ouisse C, Sebille V, Reignier J. Impact of targeted hypothermia in expanded-criteria organ donors on recipient kidney-graft function: study protocol for a multicentre randomised controlled trial (HYPOREME). BMJ Open. 2022 Mar 28;12(3):e052845. doi: 10.1136/bmjopen-2021-052845. PMID 35351701